CLINICAL TRIAL: NCT06504095
Title: The Effect of Flipped Classroom Teaching Method on Medical Error Tendency of Intern Nurses
Brief Title: The Effect of Flipped Classroom Teaching Method on Medical Error Tendencies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, NESRİN OĞURLU, Lecturer- PhD, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Medical error tendency
Record Dates: First submitted 2024-02-08; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Nursing Students; Education
Keywords: Flipped Classroom Teaching; medical error; intern nurses; nursing education

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study. It was planned to divide the students into two groups as experimental and control groups. Simple random sampling method will be used to determine the experimental and control groups. To ensure randomization, each student will be numbered and data sets (experiment and control) will be created.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Flipped Teaching Method Group) (Experimental): "The Flipped Teaching method will be used to provide patient safety training to the intervention group of students."
  Interventions: Other: intervention group (Flipped Teaching Method Group)
- Control group (Traditional Method Group) (No Intervention): "The control group of students will receive patient safety training using the traditional method. No intervention will be applied."

INTERVENTIONS:
Other: intervention group (Flipped Teaching Method Group) — "Patient safety training will be provided to students using the flipped classroom teaching method, consisting of both out-of-class and in-class activities.
  Out-of-Class Activity: For the Flipped Teaching method, a Learning Management System-Web-Based Distance Education System will be established. Lecture videos for each lesson will be uploaded to the system 7 days before the class day. Students will have the flexibility to watch the instructional videos as many times as they wish until the class day.
  In-Class Activity: The researcher will come prepared for in-class activities such as "question-answer sessions, discussions, brainstorming." No lecturing will be done by the researcher. The researcher will solely guide the students."
  Arms: intervention group (Flipped Teaching Method Group)

SUMMARY:
This study aimed to determine the effect of the flipped classroom teaching method on the medical error tendencies of intern nurses.

DETAILED DESCRIPTION:
"The World Health Organization (WHO) defines patient safety as efforts to minimize preventable harm that may occur during a patient's interaction with healthcare services. Patient safety encompasses all areas, from accurate and effective medications to safe injections, surgical procedures, and standards in other invasive procedures. Medical errors, which pose a significant risk to patient safety, have become a multidimensional issue, leading to accidents and deaths, and raising ethical-legal issues.

While there are different definitions of medical errors in the literature, the Joint Commission of Accreditation of Healthcare Organizations defines a medical error as "inappropriate and unethical behavior by a healthcare professional, resulting in harm to the patient due to inadequate and negligent behavior in professional practices."

Medical errors made by healthcare workers are a major cause of mortality and morbidity in hospitalized patients. Nurses, being the healthcare professionals who spend the longest and most continuous time with patients in the delivery of healthcare services, play a crucial role in ensuring patient safety. Teaching safe patient care is a fundamental element of nursing education. The knowledge and experiences gained during nursing education impact students' competence in ensuring and improving patient safety in their caregiving practices. Insufficient skill training and the learning process are major contributors to medical errors.

Nursing students who do not learn and experience basic nursing skills adequately may pose a risk of harm to the patients they care for. Students lacking clinical experience are at a higher risk of making unwanted errors in patient care. Therefore, it is important to increase the knowledge and awareness of nursing students regarding medical errors throughout their education.

Comprising complementary theoretical and practical sections, nursing education aims to provide students with fundamental knowledge, skills, and attitudes in the cognitive, affective, and psychomotor domains. Today's students, predominantly from Generation Y and Z, exhibit advanced thinking and quick information acquisition processes. They are willing to embrace change and constantly seek new approaches. Technology is a symbol of many aspects of their lives, and these generations are considered superior to Generation X in terms of technology use.

Educational organizations emphasize the need for nursing educators to train more competent nurses. Studies suggest that traditional teaching methods do not allow nurses to fulfill their expected responsibilities. The flipped classroom teaching method, combining the advantages of both traditional and web-based learning, encourages active learning, and enhances student performance. It reverses the traditional flow of learning, allowing students to learn the material that the instructor would traditionally present in the classroom outside of class hours through electronic materials. In-class time is then used for discussion of the material and reinforcement exercises to deepen and strengthen learning.

Students complete the relatively easy first steps, such as listening to the lecture, on their own at home. Difficult and complex applications related to higher-level steps are performed in the classroom, using active learning methods under the guidance of the instructor. This approach helps students develop critical thinking skills, learn the subject, reason, and apply current research results.

Both international and national organizations emphasize the need for nursing educators to train more competent nurses. Studies suggest that the traditional teaching method does not allow nurses to fulfill their expected responsibilities, while the flipped classroom teaching method could be a useful method for students to learn basic concepts and increase motivation and success.

Despite the challenges posed by the COVID-19 pandemic, there is a need to impart certain skills to future nurses, address the increase in the number of students, and adapt nursing education to the realities of Generation Y and Z students. Nursing education today prioritizes student-centered education and learning. The use of new methods and models in education is necessary, especially given the increasing number of students and limited resources in our country.

Requirements and conditions necessitate the exploration and implementation of new models such as flipped learning in nursing education; therefore, this research has been decided to be conducted. This study aims to determine the impact of the flipped classroom learning method on the medical error tendencies of intern nursing students. It is believed that the results of this study will contribute to raising awareness of potential medical errors, preventing them, and providing valuable insights for the improvement of nursing education. As the importance of patient safety increases due to the rising number of medical errors, this research is deemed necessary."

ELIGIBILITY:
Inclusion Criteria:

* "To be enrolled for the first time in the Nursing Care Management Course,
* To have sufficient internet access,
* To be willing to participate in the research."

Exclusion Criteria:

* To be a high school, associate, or bachelor's degree graduate in a health-related field,
* To have previously taken a course related to patient safety,
* To be unwilling to participate in the research."

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
"Determination of students' tendency towards medical errors [To be determined at the end of the study (4 weeks later)]" | To be measured at the end of the study (4 weeks later)
  "The 'Medical Error Proneness Scale', developed to measure the tendency towards medical errors, will be applied to both the experimental and control group students.. Determining and comparing the medical error proneness levels of the experimental and control groups."

CONTACTS AND LOCATIONS:
Overall Officials: NESRİN OĞURLU, Lecturer-PhD, Principal Investigator — Aydın Adnan Menderes University Aydın Vocational School of Health Services; GÜLENGÜN TÜRK, Prof.Dr., Study Director — Aydın Adnan Menderes University Faculty of Nursing, Department of Nursing Fundamentals

IPD SHARING:
Plan to Share IPD: Undecided